CLINICAL TRIAL: NCT06122285
Title: Effectiveness and Safety of Bulevirtide (BLV) Therapy in Patients With Chronic Hepatitis Delta (CHD) in Italy: a Multicenter Prospective Real Life Data Study
Brief Title: Effectiveness and Safety of Bulevirtide (BLV) Therapy in Patients With Chronic Hepatitis Delta (CHD) in Italy (D-SHIELD)
Acronym: D-SHIELD
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 184853
Record Dates: First submitted 2023-10-30; First posted 2023-11-08 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Hepatitis D
MeSH Terms: conditions — Hepatitis D | interventions — bulevirtide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hepatis Delta: Bulevirtide (BLV) at a dose of 2 mg/day subcutaneously
  Interventions: Drug: Bulevirtide

INTERVENTIONS:
Drug: Bulevirtide — dose of 2 mg/day subcutaneously

SUMMARY:
Multicenter pharmacological observational prospective, no-profit, study.

This study was designed to get a "real-life" snapshot across several Italian Hepatology centers. All HDV patients are followed up according to EASL 2017 guidelines. This allows uniformity on the indication for antiviral treatment and management of that antiviral therapy. No off-label medications are used. All data are retrievable from the patient's medical record. In addition, clinical and biochemical data from patients at month 0, 1, 2, 4, 6 and 12 of treatment, and otherwise within the study period, will be collected longitudinally.

The primary objective of the study is to describe the virological response to BLV in all patients starting BLV therapy for CHD, defined as a >2 Log decline in HDV-RNA or undetectable HDV-RNA (using the Robogene 2.0 quantitative kit, LLQ <6 IU/ml) at month 12 of therapy.

HDV patients who will start therapy with BLV 2 mg/day from May 2023, according to AIFA guidelines, will be consecutively enrolled.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Chronic hepatitis delta
* Compensated cirrhosis HDV related
* Patients who will start therapy with BLV 2 mg/day from May 2023

Exclusion Criteria:

* HDV-related decompensated cirrhosis (CPT ≥7)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with CHD (quantifiable HDV-RNA) who will start treatment with BLV 2 mg/day during the study period at the S.C. Gastroenterology and Hepatology (Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico) and at participating centers, and who met the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Describe the virological response to BLV in all patients starting BLV therapy for CHD | Month 6
  Percentage of patients with undetectable HDV RNA
Describe the virological response to BLV in all patients starting BLV therapy for CHD | Month 12
  Percentage of patients with ≥ 2 log IU/ml decline of HDV RNA

SECONDARY OUTCOMES:
Evaluation of the proportion of patients with virological response, defined as a >2 Log decline in HDV-RNA | Month 6
  Proportion of patients with virological response, defined as a >2 Log decline in HDV-RNA
Evaluation of the proportion of patients with virological response, defined as a >2 Log decline in HDV-RNA | Month 12
  Proportion of patients with virological response, defined as a >2 Log decline in HDV-RNA
Evaluation of the proportion of patients with virological response, defined as undetectable HDV-RNA | Month 6
  Proportion of patients with virological response, defined as undetectable HDV-RNA
Evaluation of the proportion of patients with virological response, defined as undetectable HDV-RNA | Month 12
  Proportion of patients with virological response, defined as undetectable HDV-RNA
Evaluation of the percentage of patients with >2 Log decrease in HDV-RNA along with normalization of ALT | Month 6
  Percentage of patients with >2 Log decrease in HDV-RNA along with normalization of ALT
Evaluation of the percentage of patients with >2 Log decrease in HDV-RNA along with normalization of ALT | Month 12
  Percentage of patients with >2 Log decrease in HDV-RNA along with normalization of ALT
Evaluation of the percentage of patients with normal ALT | Month 6
  Percentage of patients with normal ALT
Evaluation of the percentage of patients with normal ALT | Month 12
  Percentage of patients with normal ALT
Evaluation of the percentage of patients with clinical response, i.e., the percentage of patients who remain free of liver complications, such as HCC or decompensation | Month 6
  Percentage of patients who remain free of liver complications (de novo HCC or onset of decompensation)
Evaluation of the percentage of patients with clinical response, i.e., the percentage of patients who remain free of liver complications, such as HCC or decompensation | Month 12
  Percentage of patients who remain free of liver complications (de novo HCC or onset of decompensation)
Investigation of changes over time in serum levels of HBsAg (UI/mL) | Month 6
  Change in serum levels of HBsAg- by medians and ranges
Investigation of changes over time in serum levels of HBsAg (UI/mL) | Month 12
  Change in serum levels of HBsAg- by medians and ranges
Investigation of changes over time in serum levels of albumin (g/dL) | Month 6
  Change in serum levels albumin- by medians and ranges
Investigation of changes over time in serum levels of albumin (g/dL) | Month 12
  Change in serum levels albumin- by medians and ranges
Investigation of changes over time in serum levels of platelets (10e9/L) | Month 6
  Change in serum levels of platelets - by medians and ranges
Investigation of changes over time in serum levels of platelets (10e9/L) | Month 12
  Change in serum levels of platelets - by medians and ranges
Investigation of changes over time in serum levels of AFP (µg/L) | Month 6
  Change in serum levels of AFP - by medians and ranges
Investigation of changes over time in serum levels of AFP (µg/L) | Month 12
  Change in serum levels of AFP - by medians and ranges
Evaluation of treatment safety | Month 6
  Occurrence of change in serum bile acid levels (µmol/L)
Evaluation of treatment safety | Month 6
  Occurrence of adverse events
Evaluation of treatment safety | Month 12
  Occurrence of change in serum bile acid levels (µmol/L)
Evaluation of treatment safety | Month 12
  Occurrence of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation IRCCS Ca' Granda Ospedale Maggiore Policlinico, Division of Gastroenterology and Hepatology, Milan, Italy., Milan, MI, Italy